CLINICAL TRIAL: NCT01120691
Title: A 64-week Treatment, Multi-center, Randomized, Double-blind, Parallel-group, Active Controlled Study to Evaluate the Effect of QVA149 (110/50 μg o.d.) vs NVA237 (50 μg o.d.) and Open-label Tiotropium (18 μg o.d.) on COPD Exacerbations in Patients With Severe to Very Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effect of QVA149 Versus NVA237 and Tiotropium on Chronic Obstructive Pulmonary Disorder (COPD) Exacerbations
Acronym: SPARK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVA149A2304; 2009-013256-69 (EudraCT Number)
Record Dates: First submitted 2010-05-05; First posted 2010-05-11 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: QVA149; NVA237; COPD; exacerbation; combination bronchodilator
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; Glycopyrrolate; Tiotropium Bromide; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- QVA149 (Experimental): QVA149 110/50 μg capsules for inhalation, once daily delivered via Novartis Single Dose Dry Powder Inhaler (SDDPI) for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks). Salbutamol/albuterol was available for rescue medication use throughout the study.
  Interventions: Drug: QVA149; Drug: Salbutamol/albuterol
- NVA237 (Active Comparator): NVA237 50 μg capsules for inhalation, once daily delivered via Novartis Single Dose Dry Powder Inhaler (SDDPI) for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks). Salbutamol/albuterol was available for rescue medication use throughout the study.
  Interventions: Drug: NVA237; Drug: Salbutamol/albuterol
- open-label tiotropium (Active Comparator): Open-label tiotropium bromide 18 μg capsules for inhalation once daily delivered via HandiHaler® device for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks). Salbutamol/albuterol was available for rescue medication use throughout the study.
  Interventions: Drug: tiotropium; Drug: Salbutamol/albuterol

INTERVENTIONS:
Drug: QVA149 — QVA149 110/50 μg capsules for inhalation, once daily delivered via Novartis Single Dose Dry Powder Inhaler (SDDPI) for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks).
  Arms: QVA149
Drug: NVA237 — NVA237 50 μg capsules for inhalation, once daily delivered via Novartis Single Dose Dry Powder Inhaler (SDDPI) for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks).
  Arms: NVA237
Drug: tiotropium — Open-label tiotropium bromide 18 μg capsules for inhalation once daily delivered via HandiHaler® device for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks).
  Arms: open-label tiotropium
Drug: Salbutamol/albuterol — As needed throughout the study

SUMMARY:
This study is designed to assess the effect of once-daily QVA149 on COPD exacerbations in patients with severe to very severe COPD.

ELIGIBILITY:
Inclusion Criteria :

1. Male or female adults aged ≥40 years, who had signed an informed consent form prior to initiation of any study-related procedure.
2. Patients with severe to very severe Chronic Obstructive Pulmonary Disease COPD (Stage III or IV) according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines 2008.
3. Current or ex-smokers with a smoking history of at least 10 pack years (Ten pack-years were defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years).
4. Patients with a post-bronchodilator Forced Expiratory Volume in one second ( FEV1) <50% of the predicted normal value, and post-bronchodilator FEV1/ Forced Vital Capacity (FVC) <0.70 at Visit 2 (day -14). (Post refers to 1 h after sequential inhalation of 84 µg (or equivalent dose) of ipratropium bromide and 400 µg of salbutamol).
5. A documented history of at least 1 COPD exacerbation in the previous 12 months that required treatment with systemic glucocorticosteroids and/or antibiotics.

Exclusion Criteria:

1. Pregnant women or nursing mothers (pregnancy confirmed by positive urine pregnancy test).
2. Women of child-bearing potential
3. Patients requiring long term oxygen therapy (> 15 h a day) on a daily basis for chronic hypoxemia.
4. Patients who had a COPD exacerbation that required treatment with antibiotics, systemic steroids (oral or intravenous) or hospitalization in the 6 weeks prior to visit 1 or between visit 1 (Day -21) and Visit 3 (Day 1).
5. Patients who developed a COPD exacerbation during a period between visit 1 and 3 were ineligible but were permitted to be re-screened after a minimum of 6 weeks after the resolution of the COPD exacerbation.
6. Patients who had a respiratory tract infection within 4 weeks prior to visit 1 (Day -21)

   • Patients who developed an upper or lower respiratory tract infection during the screening period (up to visit 3 (Day 1) were not eligible, but were permitted to be re-screened 4 weeks after the resolution of the respiratory tract infection
7. Patients with concomitant pulmonary disease, e.g. pulmonary tuberculosis (unless confirmed by chest x-ray to be no longer active), clinically significant bronchiectasis, sarcoidosis, interstitial lung disorder or pulmonary hypertension.
8. Patients with lung lobectomy, or lung volume reduction or lung transplantation.
9. Patients who, in the judgment of the investigator, have a clinically relevant laboratory abnormality or a clinically significant condition such as (but not limited to):

   * Unstable ischemic heart disease, left ventricular failure, history of myocardial infarction, arrhythmia (excluding chronic stable Atrial Fibrillation (AF). Patients with such events not considered clinically significant by the investigator may be considered for inclusion in the study
   * history of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin
   * uncontrolled hypo- or hyperthyroidism, hypokalemia or hyper adrenergic state
   * narrow-angle glaucoma
   * Symptomatic prostatic hyperplasia or bladder-neck obstruction or moderate to severe renal impairment or urinary retention. (Patients with a Transurethral Resection of Prostate (TURP) were excluded from the study. Patients who underwent full re-section of the prostate could be considered for the study, as well as patients who were asymptomatic and stable on pharmacological treatment for the condition).
   * any condition which might have compromised patient safety or compliance, interfered with evaluation, or precluded completion of the study
10. Patients with any history of asthma indicated by (but not limited to) a blood eosinophil count > 600/mm3 (at visit 2), or onset of symptoms prior to 40 years. Patients without asthma were excluded if their eosinophil count was >600/mm3 at visit 2.
11. Patients with allergic rhinitis who used H1 antagonists or intranasal corticosteroids intermittently (treatment with a constant dose was permitted).
12. Patients with eczema (atopic), known high immunoglobulin E (IgE) levels or a known positive skin prick test in the last 5 years.
13. Patients with known history and diagnosis of alpha-1 antitrypsin deficiency.
14. Patients who were participating in the active phase of a supervised pulmonary rehabilitation program.
15. Patients with Type I or uncontrolled Type II diabetes.
16. Patients contraindicated for treatment with, or having a history of reactions/ hypersensitivity to any of the following inhaled drugs or drugs of a similar class or any component thereof:

    * anticholinergic agents
    * long and short acting beta-2 agonists
    * sympathomimetic amines.
17. Patients with a history of long QT syndrome or whose corrected QT interval (QTc) measured at visit 2 (Day -14) (Fridericia method) was prolonged (>450 ms for males and females) as confirmed by the central ECG assessor.
18. Patients with a clinically significant abnormality on the screening or baseline ECG who in the judgment of the investigator would be at potential risk if enrolled into the study. (These patients could not be re-screened).
19. Patients who needed treatments for COPD and allied conditions after the start of the study (visit 1)
20. Patients who needed treatments for COPD and allied conditions (e.g. allergic rhinitis) unless they had been stabilized
21. Patients taking other prohibited medications
22. Patients unable to use a dry powder inhaler (e.g. single dose dry powder inhaler (SDDPI), HandiHaler® device, or pressurized Metered Dose Inhaler (MDI) (rescue medication).
23. Patients unable to use an electronic patient diary.
24. Patients who were, in the opinion of the investigator known to be unreliable or non-compliant.
25. Patients who used other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of visit 1 (day -21), whichever was longer.
26. Patients who had live attenuated vaccination within 30 days prior to the screening visit or during the run-in period. Inactivated influenza vaccination, pneumococcal vaccination or any other inactivated vaccine was acceptable provided it was not administered within 48 hours prior to screening and randomization visits.

No additional exclusions were applied by the investigator, in order to ensure that the study population was representative of all eligible patients.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2224 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (291):
- United States (49):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Fairhope, Alabama
  - Novartis Investigative Site, Florence, Alabama
  - Novartis Investigative Site, Homewood, Alabama
  - Novartis Investigative Site, Jasper, Alabama
  - Novartis Investigative Site, Pine Bluff, Arkansas
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Palo Alto, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Couer D'Alene, Idaho
  - Novartis Investigative Site, Normal, Illinois
  - Novartis Investigative Site, River Forest, Illinois
  - Novartis Investigative Site, Florence, Kentucky
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Opelousas, Louisiana
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Fridley, Minnesota
  - Novartis Investigative Site, Ozark, Missouri
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Papillion, Nebraska
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, Great Neck, New York
  - Novartis Investigative Site, Massapequa, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Wilmington, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Beaver, Pennsylvania
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Salem, Virginia
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Green Bay, Wisconsin
- Argentina (13):
  - Novartis Investigative Site, Paraná Entre Ríos, Argentina
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, San Isidro, Buenos Aires
  - Novartis Investigative Site, Corrientes, Corrientes Province
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Mendoza, Mendoza Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
- Austria (5):
  - Novartis Investigative Site, Feldbach, Austria
  - Novartis Investigative Site, Grieskirchen, Austria
  - Novartis Investigative Site, Linz, Austria
  - Novartis Investigative Site, Salzburg, Austria
  - Novartis Investigative Site, Thalheim bei Wels, Austria
- Canada (9):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Joliette, Quebec
  - Novartis Investigative Site, Laval, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saint Romuald, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Colombia (6):
  - Novartis Investigative Site, Medellín, Colombia
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Armenia
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Medellín
- Czechia (16):
  - Novartis Investigative Site, Cvikov, Czech Republic
  - Novartis Investigative Site, Český Krumlov, Czech Republic
  - Novartis Investigative Site, Havlíčkův Brod, Czech Republic
  - Novartis Investigative Site, Jaroměř, Czech Republic
  - Novartis Investigative Site, Karlovy Vary, Czech Republic
  - Novartis Investigative Site, Kroměříž, Czech Republic
  - Novartis Investigative Site, Kutná Hora, Czech Republic
  - Novartis Investigative Site, Kyjov, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Rokycany, Czech Republic
  - Novartis Investigative Site, Strakonice, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Znojmo, Czech Republic
  - Novartis Investigative Site, Žatec, Czech Republic
- Denmark (7):
  - Novartis Investigative Site, Aalborg, Denmark
  - Novartis Investigative Site, Hellerup, Denmark
  - Novartis Investigative Site, Hvidovre, Denmark
  - Novartis Investigative Site, Roskilde, Denmark
  - Novartis Investigative Site, Silkeborg, Denmark
  - Novartis Investigative Site, Sønderborg, Denmark
  - Novartis Investigative Site, Copenhagen NV
- Estonia (3):
  - Novartis Investigative Site, Tallinn, Estonia
  - Novartis Investigative Site, Tartu, Estonia
  - Novartis Investigative Site, Tallinn
- Finland (3):
  - Novartis Investigative Site, Helsinki, Finland
  - Novartis Investigative Site, Jyväskylä, Finland
  - Novartis Investigative Site, Turku, Finland
- France (5):
  - Novartis Investigative Site, Beuvry, France
  - Novartis Investigative Site, Ferolles-Attily, France
  - Novartis Investigative Site, Bayonne
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
- Germany (40):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Dresden, Germany
  - Novartis Investigative Site, Heidelberg, Germany
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Marburg, Germany
  - Novartis Investigative Site, München, Germany
  - Novartis Investigative Site, Potsdam, Germany
  - Novartis Investigative Site, Teterow, Germany
  - Novartis Investigative Site, Koblenz, North Rhine-Westphalia
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düren
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freudenberg
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Gummersbach
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Langenfeld
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Oranienburg
  - Novartis Investigative Site, Radebeul
  - Novartis Investigative Site, Reinfeld
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Schwerte
  - Novartis Investigative Site, Schwetzingen
  - Novartis Investigative Site, Solingen
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Wissen
- Greece (4):
  - Novartis Investigative Site, Larissa, Greece
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Athens - GR
  - Novartis Investigative Site, Thessaloniki
- Hungary (11):
  - Novartis Investigative Site, Cegléd, Hungary
  - Novartis Investigative Site, Debrecen, Hungary
  - Novartis Investigative Site, Szarvas, Hungary
  - Novartis Investigative Site, Baja
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Deszk
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Makó
  - Novartis Investigative Site, Mosonmagyaróvár
  - Novartis Investigative Site, Sopron
  - Novartis Investigative Site, Szekszárd
- India (12):
  - Novartis Investigative Site, Hyderabad, A.p.
  - Novartis Investigative Site, Hyderbabd, Andhra Pradesh
  - Novartis Investigative Site, Nagpur - Maharastra, India
  - Novartis Investigative Site, Trivandrum, India
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Panjim
  - Novartis Investigative Site, Secunderabad
- Ireland (2):
  - Novartis Investigative Site, Dublin, Ireland
  - Novartis Investigative Site, Dublin
- Israel (8):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Italy (16):
  - Novartis Investigative Site, Osimo, AN
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Arenzano, GE
  - Novartis Investigative Site, Pisa, Italy
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Abano Terme, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Riccione, RN
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Pietra Ligure, SV
  - Novartis Investigative Site, Montecchio Maggiore, VI
- Mexico (5):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Zapopan, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
- Netherlands (13):
  - Novartis Investigative Site, Almelo, Netherlands
  - Novartis Investigative Site, Breda, Netherlands
  - Novartis Investigative Site, Enschede, Netherlands
  - Novartis Investigative Site, Harderwijk, Netherlands
  - Novartis Investigative Site, Helmond, Netherlands
  - Novartis Investigative Site, Dordrecht
  - Novartis Investigative Site, Drachten
  - Novartis Investigative Site, Hoofddorp
  - Novartis Investigative Site, Hoorn
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Roermond
  - Novartis Investigative Site, Veldhoven
  - Novartis Investigative Site, Voorburg
- Peru (6):
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Martín de Porres, Lima region
  - Novartis Investigative Site, San Miguel, Lima region
  - Novartis Investigative Site, Santiago de Surco, Lima region
- Philippines (5):
  - Novartis Investigative Site, Quezon City, National Capital Region
  - Novartis Investigative Site, Bulacan, Philippines
  - Novartis Investigative Site, Las Piñas
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Poland (6):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Mrozy
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, Humacao, Puerto Rico
- Russia (11):
  - Novartis Investigative Site, Kazan', Tatarstan Republic
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (9):
  - Novartis Investigative Site, Banská Bystrica, Slovak Republic
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Humenné, Slovak Republic
  - Novartis Investigative Site, Partizánske, Slovak Republic
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Kráľovský Chlmec, Slovakia
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Prešov, Slovakia
  - Novartis Investigative Site, Trnava, Slovakia
- South Africa (3):
  - Novartis Investigative Site, Durban, South Africa
  - Novartis Investigative Site, Newtown, Johannesburg
  - Novartis Investigative Site, Pretoria
- Spain (5):
  - Novartis Investigative Site, Alicante, Alicante
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Valencia, Valencia
- United Kingdom (18):
  - Novartis Investigative Site, Stockton, Cleveland
  - Novartis Investigative Site, Sneinton, Nottingham
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, Chertsey, Surrey
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, Gillingham
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Hereford
  - Novartis Investigative Site, Huntingdon
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Merseyside
  - Novartis Investigative Site, Portsmouth
  - Novartis Investigative Site, Telford
  - Novartis Investigative Site, Wolverhampton

REFERENCES:
- [Derived] Wedzicha JA, Decramer M, Ficker JH, Niewoehner DE, Sandstrom T, Taylor AF, D'Andrea P, Arrasate C, Chen H, Banerji D. Analysis of chronic obstructive pulmonary disease exacerbations with the dual bronchodilator QVA149 compared with glycopyrronium and tiotropium (SPARK): a randomised, double-blind, parallel-group study. Lancet Respir Med. 2013 May;1(3):199-209. doi: 10.1016/S2213-2600(13)70052-3. Epub 2013 Apr 23. PMID 24429126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 3865 participants were screened of whom 2224 were randomized to 1 of the 3 treatment groups (QVA149, NVA237 or tiotropium) in a 1:1:1 ratio for at least 64 weeks (maximum 76 weeks) of treatment period.
Pre-assignment Details: 5 (QVA149), 2 (NVA237) and 3 (tiotropium) participants were randomized but did not receive study drug.
Groups:
- QVA149: QVA149 110/50 μg capsules for inhalation, once daily delivered via Novartis Single Dose Dry Powder Inhaler (SDDPI) for at least 64 weeks of double blind treatment period. Salbutamol/albuterol was available for rescue medication use throughout the study.
- NVA237: NVA237 50 μg capsules for inhalation, once daily delivered via Novartis Single Dose Dry Powder Inhaler (SDDPI) for at least 64 weeks of double blind treatment period. Salbutamol/albuterol was available for rescue medication use throughout the study.
Period: Overall Study
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Started | 741 | 741 | 742
Full Analysis Set (FAS) | 736 | 739 | 739
Safety Set (SAF) | 736 | 740 | 739
Modified Safety Set (mSAF) | 729 | 740 | 737
Modified Full Analysis Set (mFAS) | 729 | 739 | 737
Completed | 570 | 538 | 559
Not Completed | 171 | 203 | 183
Not completed — Adverse Event | 59 | 67 | 47
Not completed — Subject withdrew consent | 33 | 50 | 44
Not completed — Death | 21 | 22 | 24
Not completed — Unsatisfactory therapeutic effect | 18 | 32 | 38
Not completed — Administrative problems | 15 | 8 | 9
Not completed — Protocol deviation | 13 | 12 | 12
Not completed — Lost to Follow-up | 5 | 6 | 4
Not completed — Abnormal test procedure result(s) | 3 | 2 | 1
Not completed — Patient's inability to use the device | 3 | 1 | 0
Not completed — Abnormal laboratory value(s) | 1 | 3 | 4

BASELINE CHARACTERISTICS:
Population: The modified safety set (mSAF set) includes all patients in the safety set except patients from a site who had major GCP issues.
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium | Total
Number analyzed (Participants) | 729 | 740 | 737 | 2206
Age Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.07) | 63.1 (7.98) | 63.6 (7.79) | 63.3 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 198 | 184 | 555
  Male | 556 | 542 | 553 | 1651

OUTCOME MEASURES:

1. Primary Outcome: Rate of Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations in QVA149 and NVA237 Treatment Arms During the Treatment Period.
Description: A Chronic Obstructive Pulmonary Disease (COPD) exacerbation was defined as a worsening of two or more of the following major symptoms for at least 2 consecutive days: dyspnea, sputum volume or sputum purulence OR a worsening of any 1 major symptom together with an increase in any 1 of the following minor symptoms for at least 2 consecutive days: sore throat, colds (nasal discharge and/or nasal congestion), fever without other cause, cough or wheezing. A COPD exacerbation was considered of moderate severity if treatment with systemic glucocorticosteroids or antibiotics or both was required and severe if hospitalization was required. An emergency room (ER) visit of longer than 24 hours was considered a hospitalization.
  Rate of moderate or severe exacerbations per year = total number of moderate or severe exacerbations / total number of treatment years
Time Frame: 64 weeks
Population: Modified Full Analysis Set (mFAS) included all patients in the Full analysis set except patients from a site , which had major issues with Good Clinical Practice (GCP) compliance.
Measure: Number; unit: Exacerbations per year
Units Other Than Participants: Moderate to Severe COPD Exacerbation
Groups:
- QVA149: QVA149 : QVA149 110/50 μg capsules for inhalation, once daily delivered via Novartis Single Dose Dry Powder Inhaler (SDDPI) for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks). Salbutamol/albuterol was available for rescue medication use throughout the study.
- NVA237: NVA237 : NVA237 50 μg capsules for inhalation, once daily delivered via Novartis Single Dose Dry Powder Inhaler (SDDPI) for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks). Salbutamol/albuterol was available for rescue medication use throughout the study.
Arm/Group | QVA149 | NVA237
Number analyzed (Participants) | 729 | 739
Number analyzed (Moderate to Severe COPD Exacerbation) | 812 | 900
Exacerbations per year | 0.94 | 1.07

2. Secondary Outcome: Rate of Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations in QVA149 and Open-label Tiotropium Treatment Arms During the Treatment Period.
Description: as for outcome 1
Time Frame: 76 weeks
Population: Modified Full Analysis Set (mFAS) included all patients in the Full analysis set except patients from a site, which had major issues with GCP compliance.
Measure: Number; unit: Exacerbations per year
Units Other Than Participants: Moderate to Severe COPD Exacerbation
Arm/Group | QVA149 | Open-label Tiotropium
Number analyzed (Participants) | 729 | 737
Number analyzed (Moderate to Severe COPD Exacerbation) | 812 | 898
Exacerbations per year | 0.94 | 1.06

3. Secondary Outcome: Time to First Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Between QVA149, NVA237 and Open Label Tiotropium During the Treatment Period
Description: as for outcome 1
Time Frame: 64 weeks
Population: Modified Full Analysis Set (mFAS) included all patients in the Full analysis set except patients from a site, which had major issues with GCP compliance. Only patients with a moderate or severe COPD exacerbation were included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- QVA149: QVA149 : QVA149 110/50 μg capsules for inhalation, once daily delivered via Novartis Single Dose Dry Powder Inhaler (SDDPI)for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks). Salbutamol/albuterol was available for rescue medication use throughout the study.
- NVA237: NVA237 : NVA237 50 μg capsules for inhalation, once daily delivered via Novartis Single Dose Dry Powder Inhaler (SDDPI)for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks). Salbutamol/albuterol was available for rescue medication use throughout the study.
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Number analyzed (Participants) | 419 | 426 | 402
days | 296 [267 to 358] | 287 [255 to 325] | 331 [280 to 390]

4. Secondary Outcome: Rate of Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations Requiring the Use of Both Systemic Glucocorticosteroids and Antibiotics
Description: Rate of moderate or severe exacerbations per year = total number of moderate or severe exacerbations / total number of treatment years
Time Frame: 64 weeks
Population: Modified Full Analysis Set (mFAS) included all patients in the Full analysis set except patients from a site, which had major issues with GCP compliance. The Full Analysis Set (FAS) includes all randomized patients who received at least one dose of study drug and data was available for analysis.
Measure: Number; unit: exacerbations per year
Units Other Than Participants: exacerbations
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Number analyzed (Participants) | 729 | 739 | 737
Number analyzed (exacerbations) | 403 | 491 | 461
exacerbations per year | 0.46 | 0.58 | 0.54

5. Secondary Outcome: Number of Days With Moderate or Severe Exacerbation That Required Treatment With Systemic Corticosteroids and Antibiotics
Description: The number of exacerbation days is defined as the sum of the duration of days recorded as an exacerbation for all exacerbations recorded per patient.
Time Frame: 64 weeks
Population: Modified Full Analysis Set (mFAS) included all patients in the Full analysis set except patients from a site with GCP non-compliance. This is a sub-group analysis with mutually exclusive population in each category for analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Number analyzed (Participants) | 528 | 575 | 556
Days
  systemic corticosteroids [n= 97, 108, 109] | 20.49 (25.426) | 25.22 (42.674) | 17.57 (17.797)
  antibiotics [n= 195, 177, 177] | 25.08 (47.035) | 18.10 (21.790) | 25.94 (50.007)
  corticosteroids and antibiotic [n= 266, 290, 270] | 22.10 (49.999) | 26.18 (52.336) | 22.03 (42.513)

6. Secondary Outcome: Time to Study Withdrawal or Premature Discontinuation for Any Reason Between QVA149 (110/50 µg q.d.), NVA237 (50 µg q.d.) and Open Label Tiotropium (18 µg q.d.) During the Treatment Period.
Description: Time to Study Withdrawal or Premature Discontinuation for Any Reason was analyzed for each treatment group using a Kaplan-Meier estimation for the modified safety set. Patients who did not discontinue early were censored at the final visit of the treatment phase.
Time Frame: 64 weeks
Population: Modified safety set (mSAF set) includes all patients in the safety set except patients from a site who had major GCP issues. The Safety set includes all patients who received at least one dose of study drug whether or not being randomized. Analysis population included patients with study withdrawal or premature discontinuation for any reason.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Number analyzed (Participants) | 159 | 202 | 178
days | NA [NA to NA] — Less than 50% of patients had withdrawn from the study or prematurely discontinued for any reason. | NA [NA to NA] — Less than 50% of patients had withdrawn from the study or prematurely discontinued for any reason. | NA [NA to NA] — Less than 50% of patients had withdrawn from the study or prematurely discontinued for any reason.

7. Secondary Outcome: Percentage of Patients With Study Withdrawal or Premature Discontinuation for Any Reason Between QVA149 (110/50 µg q.d.), NVA237 (50 µg q.d.) and Open Label Tiotropium (18 µg q.d.)During the Treatment Period
Description: Percentage of Patients With Study Withdrawal or Premature Discontinuation for Any Reason was analyzed for each treatment group using a Kaplan-Meier estimation for the modified safety set. Patients who did not discontinue early were censored at the final visit of the treatment phase.
Time Frame: 64 weeks
Population: Modified safety set (mSAF set) includes all patients in the safety set except patients from a site who had major GCP issues. The Safety set includes all patients who received at least one dose of study drug whether or not being randomized
Measure: Number; unit: percentage of participants
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Number analyzed (Participants) | 729 | 740 | 737
percentage of participants | 21.8 | 27.3 | 24.2

8. Secondary Outcome: Cumulative Rates of Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations for Multiple COPD Exacerbation at Different Time Points
Description: Cumulative rates were estimated using Anderson and Gill method. Chronic Obstructive Pulmonary Disease (COPD) exacerbations are considered to be moderate if treatment with systemic corticosteroids and/or antibiotics was required. COPD exacerbations are considered to be severe if treatment for moderate severity and hospitalization were required. Rate of moderate or severe exacerbations per year = total number of moderate or severe exacerbations / total number of treatment years
Time Frame: 26, 52, 64, 76 weeks
Population: Modified Full Analysis Set(mFAS) included all patients in the Full Analysis Set (FAS) except patients from a site, which had major issues with GCP compliance. FAS include all randomized patients who received at least one dose of study drug and data was available for analysis.
Measure: Number (95% Confidence Interval); unit: exacerbations per year
Units Other Than Participants: Moderate or Severe COPD Exacerbations
Groups:
- Open-label Tiotropium: Open-label tiotropium bromide 18 μg capsules for inhalation once daily delivered via HandiHaler® device for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks.Salbutamol/albuterol was available for rescue medication use throughout the study.
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Number analyzed (Participants) | 729 | 739 | 737
Number analyzed (Moderate or Severe COPD Exacerbations) | 831 | 926 | 897
exacerbations per year
  26 weeks | 0.57 [0.51 to 0.62] | 0.65 [0.58 to 0.71] | 0.63 [0.56 to 0.70]
  52 weeks | 0.99 [0.91 to 1.09] | 1.13 [1.03 to 1.25] | 1.11 [1.00 to 1.23]
  64 weeks | 1.19 [1.08 to 1.30] | 1.36 [1.24 to 1.49] | 1.31 [1.19 to 1.46]
  76 weeks | 1.39 [1.27 to 1.53] | 1.59 [1.45 to 1.74] | 1.55 [1.40 to 1.71]

9. Secondary Outcome: Pre-dose Forced Expiratory Volume in 1 Second (FEV-1) After 4, 12, 26, 38, 52 and 64 Weeks of Treatment Between QVA149, NVA237 and Open Label Tiotropium
Description: Pulmonary function assessments were performed using centralized spirometry. The spirometer was customized and programmed according to the requirements of the study protocol in accordance with American Thoracic Society (ATS) standards.
  Spirometry measurements taken were FEV1 at -45 minutes and -15 minutes pre-dose. Three acceptable maneuvers had to be performed for each time point. The FEV1 values recorded had to be the highest values measured irrespective of whether or not they occurred on the same curve.
  The mixed model for analysis contained treatment as a fixed effect with average of the 45 minutes and 15 minutes pre dose FEV1 measurements at day 1 as the baseline measurement, FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at -14 Day) as covariates.
Time Frame: 4, 12, 26, 38, 52 and 64 weeks
Population: Modified Full Analysis Set(mFAS) included all patients in the Full Analysis Set (FAS) except patients from a site, which had major issues with GCP compliance. FAS include all randomized patients who received at least one dose of study drug and data was available for analysis. Each category has patients with assessable data at that particular time.
Measure: Least Squares Mean (Standard Error); unit: L (liters)
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Number analyzed (Participants) | 729 | 739 | 737
L (liters)
  predose FEV1 Week 4 (n= 656,654,630) | 1.08 (0.009) | 0.99 (0.009) | 1.00 (0.009)
  predose FEV1 Week 12 (n= 666,663,653) | 1.08 (0.010) | 1.01 (0.009) | 1.01 (0.009)
  predose FEV1 Week 26 (n= 604,577,599) | 1.07 (0.010) | 0.99 (0.010) | 1.00 (0.010)
  predose FEV1 Week 38 (n= 593,549,583) | 1.08 (0.011) | 1.00 (0.011) | 1.00 (0.011)
  predose FEV1 Week 52 (n= 557,538,548) | 1.05 (0.011) | 0.98 (0.011) | 0.99 (0.011)
  predose FEV1 Week 64 (n= 549,504,530) | 1.05 (0.011) | 0.98 (0.011) | 0.99 (0.011)

10. Secondary Outcome: Pre-dose Forced Vital Capacity (FVC)After 4, 12, 26, 38, 52 and 64 Weeks of Treatment Between QVA149, NVA237 and Open Label Tiotropium
Description: Pulmonary function assessments were performed using centralized spirometry. The spirometer was customized and programmed according to the requirements of the study protocol in accordance with American Thoracic Society (ATS) standards.
  Pre-dose Forced Vital Capacity (FVC) is defined as the average of the -15 minutes and the -45 minutes FVC values. Baseline is defined as the average of the -45 minutes and -15 minutes FVC values taken on day 1 prior to first dose. FVC data taken within 6h of rescue medication or within 7 days of systemic corticosteroid is excluded from this analysis
Time Frame: 4, 12, 26, 38, 52 and 64 weeks
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: L (liters)
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Number analyzed (Participants) | 729 | 739 | 737
L (liters)
  predose FVC Week 4 (n= 656,654,630) | 2.74 (0.020) | 2.59 (0.019) | 2.60 (0.019)
  predose FVC Week 12 (n= 623,621,619) | 2.77 (0.021) | 2.63 (0.021) | 2.65 (0.021)
  predose FVC Week 26 (n= 604,577,599) | 2.73 (0.023) | 2.60 (0.022) | 2.61 (0.022)
  predose FVC Week 38 (n= 592,548,580) | 2.76 (0.025) | 2.65 (0.025) | 2.63 (0.025)
  predose FVC Week 52 (n= 557,538,547) | 2.68 (0.025) | 2.58 (0.025) | 2.58 (0.025)
  predose FVC Week 64 (n= 549,502,526) | 2.67 (0.025) | 2.57 (0.025) | 2.59 (0.025)

11. Secondary Outcome: Change in Mean Daily Use (Number of Puffs) of Rescue Therapy Between QVA149, NVA237 and Open Label Tiotropium From Baseling Over the 64 Week Treatment Period
Description: The severe or less FEV1 % predicted (post bronchodilator)>=30%; very severe=> FEV1 % predicted(the post bronchodilator)<30%.Number of puffs of rescue medication taken in the previous 12 hours was recorded in patient diary in the morning and in the evening for 26 weeks.The total number of puffs per day was calculated and divided by the number of days with data to determine the mean daily number of puffs of rescue medication for each patient.Rescue medication data recorded during the 14 day run-in was used to calculate the baseline.A negative change from baseline indicates improvement. A mixed model was used with treatment as a fixed effect with baseline number of puffs and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates.
Time Frame: Baseline (14 day run-in), 64 weeks
Population: Modified Full Analysis Set mFAS included all patients in the Full analysis set except patients from a site,which had major issues with GCP compliance. The Full Analysis Set includes all randomized patients who received at least one dose of study drug and data was available for analysis. Patients with evaluable data were included in this analysis
Measure: Least Squares Mean (Standard Error); unit: # puffs
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Number analyzed (Participants) | 708 | 724 | 709
# puffs
  Mean Daily # puffs Severe or Less(n=565,575,561) | -2.3 (0.137) | -1.5 (0.135) | -1.6 (0.136)
  Mean Daily # puffs Very Severe (n=143,149,148) | -2.1 (0.234) | -1.1 (0.228) | -1.0 (0.228)

12. Secondary Outcome: Change From Baseline of Percentage of Days Without Rescue Therapy Use Between QVA149,NVA237 and Open Label Tiotropium Over the 64 Week Treatment Period
Description: A day with no rescue medication use is defined from the diary data as any day where the patient recorded no rescue medicine use during the previous 12 hours. The percentage of days is calculated by the number of days with no rescue medicine use/total number of days with evaluable data X 100. A mixed model was used with treatment as a fixed effect with baseline number of puffs and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: Baseline (14 day run-in), 64 weeks
Population: Modified Full Analysis Set(mFAS)included all patients in the Full analysis set except patients from a site,which had major issues with GCP compliance. The Full Analysis Set includes all randomized patients who received at least one dose of study drug and data was available for analysis. Patients with evaluable data were included in this analysis
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Number analyzed (Participants) | 701 | 720 | 703
percentage of days | 29.36 (1.445) | 21.65 (1.410) | 23.86 (1.422)

13. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Scores Between QVA149, NVA237 and Open Label Tiotropium Over 12, 26, 38, 52 and 64 Weeks of Treatment
Description: St. George's Respiratory Questionnaire (SGRQ) is a health related quality of life questionnaire consisting of 51 items in three components: symptoms, activity, and impacts. The lowest possible value is zero and the highest 100. Higher values correspond to greater impairment in quality of life. Mixed model used baseline SGRQ, baseline inhaled corticosteroid (ICS) use, Forced Expiratory Volume in 1 Second (FEV1) prior to inhalation of short acting beta-agonist (SABA), and FEV1 45 minutes post-inhalation of SABA as covariates. SGRQ total score is the sum of the scores from the three components; symptoms, activity and impacts.
Time Frame: 12, 26, 38, 52 and 64 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Number analyzed (Participants) | 729 | 739 | 737
units on a scale
  Week 12 (n= 694,694,676) | 44.69 (0.612) | 47.13 (0.603) | 47.62 (0.607)
  Week 26 (n= 684,677,658) | 44.06 (0.655) | 45.93 (0.647) | 45.77 (0.651)
  Week 38 (n= 648,626,635) | 42.72 (0.667) | 45.53 (0.663) | 45.86 (0.660)
  Week 52 (n= 625,593,613) | 43.38 (0.722) | 45.96 (0.723) | 46.21 (0.714)
  Week 64 (n= 600,564,579) | 43.39 (0.778) | 45.46 (0.780) | 46.08 (0.778)

ADVERSE EVENTS:
Description: Modified safety set (mSAF set) includes all patients in the safety set except patients from a site who had major GCP issues. The Safety set includes all patients who received at least one dose of study drug whether or not being randomized. Analysis population included patients with study withdrawal or premature discontinuation for any reason.
Groups:
- Open-label Tiotropium: Open-label tiotropium bromide 18 μg capsules for inhalation once daily delivered via HandiHaler® device. for at least 64 weeks of double blind treatment period (study duration was up to 76 weeks). Salbutamol/albuterol was available for rescue medication use throughout the study.
Arm/Group | QVA149 | NVA237 | Open-label Tiotropium
Serious Adverse Events (participants affected / at risk) | 167/729 | 179/740 | 165/737
Other Adverse Events (participants affected / at risk) | 656/729 | 671/740 | 666/737
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=729) | NVA237 (N=740) | Open-label Tiotropium (N=737)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 4 | 2
Angina pectoris (Cardiac disorders) | 1 | 3 | 1
Angina unstable (Cardiac disorders) | 1 | 2 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 3 | 4
Atrial flutter (Cardiac disorders) | 0 | 2 | 1
Cardiac arrest (Cardiac disorders) | 1 | 4 | 2
Cardiac failure (Cardiac disorders) | 1 | 1 | 4
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 3 | 3
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 3 | 0
Cor pulmonale chronic (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 3 | 2 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 3 | 4
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 2 | 0
Congenital laryngeal stridor (Congenital, familial and genetic disorders) | 0 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal congestion (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Adverse drug reaction (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Cyst (General disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 2 | 3
Oedema peripheral (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 2
Sudden cardiac death (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0
Thrombosis in device (General disorders) | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 1 | 0
Abscess intestinal (Infections and infestations) | 1 | 0 | 0
Abscess rupture (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 2 | 5
Bronchopneumonia (Infections and infestations) | 2 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0
Haemophilus infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 4 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 14 | 24 | 13
Lower respiratory tract infection bacterial (Infections and infestations) | 2 | 5 | 1
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1 | 0
Otitis media chronic (Infections and infestations) | 1 | 0 | 0
Perineal abscess (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 23 | 25 | 24
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 1 | 0
Rabies (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 2 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 2 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 3 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 20 | 20 | 10
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 6 | 5 | 3
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Carcinoid tumour of the caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gliosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 4
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 2 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 3
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0
Movement disorder (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 3 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Bladder dysfunction (Renal and urinary disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 107 | 116 | 87
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 6
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pollution (Social circumstances) | 1 | 0 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 2
Arterial stenosis (Vascular disorders) | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 2 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Phlebitis deep (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=729) | NVA237 (N=740) | Open-label Tiotropium (N=737)
Tachycardia (Cardiac disorders) | 3 | 8 | 3
Abdominal pain (Gastrointestinal disorders) | 6 | 11 | 9
Abdominal pain upper (Gastrointestinal disorders) | 7 | 7 | 8
Constipation (Gastrointestinal disorders) | 8 | 11 | 4
Diarrhoea (Gastrointestinal disorders) | 21 | 11 | 15
Dry mouth (Gastrointestinal disorders) | 4 | 13 | 16
Dyspepsia (Gastrointestinal disorders) | 13 | 10 | 15
Gastritis (Gastrointestinal disorders) | 12 | 5 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 4 | 9
Nausea (Gastrointestinal disorders) | 9 | 12 | 4
Toothache (Gastrointestinal disorders) | 9 | 4 | 6
Fatigue (General disorders) | 4 | 8 | 3
Non-cardiac chest pain (General disorders) | 14 | 11 | 9
Oedema peripheral (General disorders) | 22 | 18 | 16
Pyrexia (General disorders) | 26 | 24 | 22
Bronchitis (Infections and infestations) | 32 | 36 | 26
Influenza (Infections and infestations) | 23 | 22 | 19
Lower respiratory tract infection (Infections and infestations) | 49 | 68 | 69
Lower respiratory tract infection bacterial (Infections and infestations) | 6 | 8 | 4
Nasopharyngitis (Infections and infestations) | 98 | 81 | 90
Oral candidiasis (Infections and infestations) | 11 | 10 | 12
Pharyngitis (Infections and infestations) | 17 | 11 | 10
Pneumonia (Infections and infestations) | 11 | 13 | 10
Rhinitis (Infections and infestations) | 9 | 10 | 6
Sinusitis (Infections and infestations) | 12 | 20 | 21
Upper respiratory tract infection (Infections and infestations) | 26 | 25 | 28
Upper respiratory tract infection bacterial (Infections and infestations) | 119 | 123 | 109
Urinary tract infection (Infections and infestations) | 27 | 19 | 15
Viral upper respiratory tract infection (Infections and infestations) | 70 | 75 | 72
Contusion (Injury, poisoning and procedural complications) | 9 | 4 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 14 | 11 | 11
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 | 4 | 7
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 12 | 9 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 10 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 33 | 36
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 9 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 9 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 8 | 5
Dizziness (Nervous system disorders) | 13 | 12 | 8
Headache (Nervous system disorders) | 30 | 33 | 39
Depression (Psychiatric disorders) | 4 | 2 | 9
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 618 | 639 | 629
Cough (Respiratory, thoracic and mediastinal disorders) | 40 | 39 | 25
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 42 | 32
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 | 32 | 29
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 7 | 13 | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 3
Hypertension (Vascular disorders) | 30 | 20 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.